CLINICAL TRIAL: NCT07347314
Title: Enfortumab Vedotin in Patients With Locally Advanced or Metastatic Small Bowel Adenocarcinoma Refractory or Intolerant to Platinum-based Combination Therapy: a Multicenter, Phase II Investigator-initiated Trial (ENVELOPE, NCCH2412/MK015)
Brief Title: Enfortumab Vedotin in Patients With Advanced Small Bowel Adenocarcinoma Refractory or Intolerant to Platinum-based Combination Therapy
Acronym: ENVELOPE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Japan (Other Government)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCH2412/MK015
Record Dates: First submitted 2025-12-22; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Advanced Small Bowel Adenocarcinoma
Keywords: enfortumab vedotin; small bowel adenocarcinoma; advanced
MeSH Terms: interventions — enfortumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enfortumab vedotin (Experimental)
  Interventions: Drug: Enfortumab vedotin

INTERVENTIONS:
Drug: Enfortumab vedotin — Enfortumab vedotin 1.25 mg/kg administered intravenously over at least 30 minutes on Days 1, 8, and 15 of each 28-day cycle, continued until disease progression, unacceptable toxicity, withdrawal of consent, or other protocol-defined discontinuation.

SUMMARY:
Small bowel adenocarcinoma is a rare cancer with a poor prognosis. For patients with locally advanced or metastatic disease, the usual first treatment is chemotherapy with platinum-based combinations such as FOLFOX or CapeOX. However, once the cancer grows after this treatment or the side effects become too severe, there is no widely accepted standard second-line therapy, and outcomes are generally poor. New treatment options are therefore urgently needed. Recent retrospective research from our group has shown that the majority of the small bowel adenocarcinomas strongly express a protein called Nectin-4 on the surface of cancer cells. High Nectin-4 expression was also associated with poorer survival, suggesting that Nectin-4 could be a crucial treatment target in this disease.

Enfortumab vedotin is a targeted anticancer drug called an antibody-drug conjugate. It combines an antibody that recognizes Nectin-4 with vedotin, a cytotoxic anticancer agent (payload). After enfortumab vedotin binds to Nectin-4 on the tumor cell surface, it is taken up into the cell and releases the anticancer payload, which damages the cell's internal structure and leads to cell death and apoptosis. Enfortumab vedotin has already shown meaningful antitumor activity and an acceptable safety profile in patients with advanced urothelial carcinoma and is approved over the world. However, its efficacy has never been formally evaluated in patients with small bowel adenocarcinoma.

ENVELOPE is a multicenter, single-arm, phase II investigator-initiated trial designed to evaluate the efficacy and safety of enfortumab vedotin in patients with locally advanced or metastatic small bowel adenocarcinoma that has progressed during or after, or is intolerant to, platinum-based combination chemotherapy (FOLFOX or CapeOX). Eligible patients are adults (aged 18 years or older) with histologically or cytologically confirmed small bowel adenocarcinoma, a good performance status, adequate organ function, and at least one measurable lesion on a CT scan. Patients who have genomic alterations that make them candidates for previously approved "tumor-agnostic" targeted drugs (for example, high microsatellite instability or high tumor mutational burden) must already have tried and not benefited from, or not tolerated, those treatments. Testing positive for Nectin-4 is not required to take part in this study.

Participants will receive enfortumab vedotin as an intravenous infusion at a dose of 1.25 mg/kg on days 1, 8, and 15 of each 28-day treatment cycle. Treatment will continue as long as the cancer does not grow and side effects remain manageable. Tumor scans with contrast-enhanced CT will be performed every 8 weeks up to week 24 and every 12 weeks thereafter to monitor the response of the enfortumab vedotin. The primary objective is to determine the proportion of patients achieving a tumor response to enfortumab vedotin, as assessed by independent radiologic review. Key secondary objectives include progression-free survival, overall survival, duration of response, and safety profiling.

In addition, this study includes a prespecified translational research program. Tumor samples will be examined for Nectin-4 expression using immunohistochemistry, and researchers will investigate the relationship between Nectin-4 levels and the effects of enfortumab vedotin. Blood and tissue samples will also be collected before treatment, during treatment, and at the time of cancer progression, when possible, for detailed "multi-omics" analyses. These translational studies aim to elucidate why some patients respond whereas others do not, and to identify biomarkers that could inform future treatment strategies for small bowel adenocarcinoma.

The ENVELOPE trial has been approved by the Institutional Review Board of the National Cancer Center, Japan, as well as by the ethics committees at participating sites. The study is funded by the Japan Agency for Medical Research and Development (AMED), and enfortumab vedotin is supplied by Astellas Pharma. Enrollment began in October 2025 and is planned to continue through October 2027, with patients followed for at least 12 months after the last participant is enrolled.

DETAILED DESCRIPTION:
Small bowel adenocarcinoma is a rare gastrointestinal malignancy that accounts for fewer than 3% of all gastrointestinal cancers and is associated with poor prognosis. Most patients are diagnosed at an advanced stage because lesions in the distal duodenum, jejunum, and ileum are difficult to detect endoscopically, and symptoms such as anemia, obstruction, or bleeding often appear only after the disease has progressed. For patients with locally advanced or metastatic small bowel adenocarcinoma, fluoropyrimidine plus oxaliplatin regimens such as FOLFOX and CapeOX are widely used as first-line systemic therapy. Prospective studies have reported objective response rates of approximately 40-50% and median overall survival of about 13-20 months with these platinum-based combinations. However, there is no established standard of care beyond first-line treatment, and outcomes after failure of platinum-based chemotherapy are dismal, with small retrospective series suggesting modest activity of regimens such as irinotecan-based chemotherapy or taxanes and very low response rates in routine practice. In the absence of targetable alterations qualifying for tumor-agnostic approved therapies, best supportive care remains the default recommendation for many patients after failure of first-line therapy.

Enfortumab vedotin is an antibody-drug conjugate composed of a fully human IgG1κ monoclonal antibody directed against the cell adhesion molecule Nectin-4, linked via a protease-cleavable linker to the microtubule inhibitor monomethyl auristatin E. Binding of enfortumab vedotin to Nectin-4 on the tumor cell surface leads to internalization of the antibody-drug conjugate and intracellular release of monomethyl auristatin E, resulting in disruption of tubulin polymerization, cell-cycle arrest at the G2/M phase, and apoptotic cell death. Non-clinical studies have shown high-affinity and selective binding to Nectin-4, Nectin-4-dependent intracellular delivery of monomethyl auristatin E, direct cytotoxicity against Nectin-4-positive tumor cells, and bystander killing of adjacent Nectin-4-negative cells. In clinical trials in patients with urothelial carcinoma, the same schedule used in this trial (1.25 mg/kg intravenously on days 1, 8, and 15 of a 28-day cycle) has demonstrated clinically meaningful antitumor activity and an acceptable safety profile in phase I-III studies, leading to regulatory approval in that indication.

There are no published clinical data for enfortumab vedotin in small bowel adenocarcinoma. To address this gap, the National Cancer Center Hospital conducted immunohistochemical analyses of Nectin-4 in tumor samples from patients with small bowel adenocarcinoma. Among 51 consecutively diagnosed cases, Nectin-4 expression was detected in 42 tumors (82.4%). In patients who received palliative chemotherapy, Nectin-4 positivity was associated with significantly shorter overall survival compared with Nectin-4-negative disease (median 12.6 vs 43.2 months), and higher levels of Nectin-4 expression tended to correlate with worse outcomes. In multivariable analysis, poor performance status and Nectin-4 positivity were both identified as independent adverse prognostic factors. These findings suggest that Nectin-4 is both highly expressed and prognostically unfavorable in small bowel adenocarcinoma, providing a strong biological rationale to investigate Nectin-4-targeted therapy in this setting.

This investigator-initiated study is a prospective, multicenter, open-label, single-arm Phase II trial designed to evaluate the antitumor activity and safety of enfortumab vedotin in adults with locally advanced or metastatic small bowel adenocarcinoma that is refractory or intolerant to platinum-based combination therapy. Eligible patients must have histologically or cytologically confirmed small bowel adenocarcinoma that is unresectable, metastatic, or recurrent after prior curative surgery, Eastern Cooperative Oncology Group performance status 0-1, at least one measurable lesion by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 on contrast-enhanced computed tomography within 14 days before registration, and prior treatment with FOLFOX or CapeOX with documented progression, recurrence, or discontinuation due to toxicity. Where prior comprehensive genomic testing has identified alterations qualifying for tumor-agnostic approved therapies (for example, high microsatellite instability or mismatch-repair deficiency, BRAF V600E mutation), patients must be refractory or intolerant to such therapies. Nectin-4 expression is not required for enrollment, in line with experience in urothelial carcinoma, where benefit has been observed regardless of Nectin-4 level. Key exclusion criteria include active or prior interstitial lung disease, poorly controlled diabetes, clinically significant ocular surface disease, and uncontrolled comorbidities that could compromise protocol therapy.

Enfortumab vedotin will be administered at a dose of 1.25 mg/kg as an intravenous infusion on days 1, 8, and 15 of each 28-day cycle. Treatment will be continued until radiographic or clinical disease progression, unacceptable toxicity, withdrawal of consent. Dose delays, interruptions, and stepwise dose reductions are specified to manage treatment-related toxicities, particularly peripheral neuropathy, skin reactions, and metabolic adverse events, based on experience from prior trials in urothelial carcinoma. Supportive care measures, including antiemetics, analgesics, nutritional support, and local radiotherapy for symptom control, are permitted according to institutional practice, while concurrent antineoplastic therapies other than the study drug are prohibited.

Tumor assessments with contrast-enhanced CT of the chest, abdomen, and pelvis will be performed every 8 weeks up to week 24 and every 12 weeks thereafter, or as clinically indicated, until documented disease progression. The best overall response and objective response rate will be evaluated according to RECIST version 1.1 by a blinded, independent central review committee, with local investigator assessments also collected for the secondary endpoint. Safety will be monitored throughout treatment and for a predefined follow-up period, with adverse events graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events. Particular attention will be paid to skin toxicity, peripheral neuropathy, hyperglycemia, and ocular events, which have been identified as important adverse drug reactions for enfortumab vedotin in other tumor types. An independent committee will periodically review accumulating safety and efficacy data to support ongoing risk-benefit evaluation.

The primary efficacy endpoint is the objective response rate based on blinded independent central review in the full analysis set. The statistical design is an exact binomial single-stage phase II design with a null hypothesis objective response rate of 5%, reflecting the limited activity of existing second-line options, and an expected objective response rate of 25% for enfortumab vedotin. With a one-sided alpha of 0.05 and 90% power, 25 evaluable patients are required; allowing for a small number of non-evaluable cases, the planned sample size is 27 patients. Secondary endpoints include investigator-assessed objective response rate, disease control rate, progression-free survival, overall survival, duration of response, time to response, and safety outcome.

A prespecified translational research program is embedded in the trial. Archival tumor tissue or a pretreatment biopsy is required for enrollment whenever feasible. Tumor Nectin-4 expression will be evaluated centrally by immunohistochemistry, and exploratory analyses will investigate the association between Nectin-4 expression levels and clinical outcomes with enfortumab vedotin. Additionally, blood and tissue biospecimens will be collected at baseline, during treatment, and at disease progression, where possible, for multi-omics analyses. These studies aim to elucidate the mechanisms of sensitivity and resistance, identify predictive and prognostic biomarkers, and generate hypotheses for subsequent biomarker-driven trials in small bowel adenocarcinoma.

The trial is conducted under the oversight of a central coordinating committee, in accordance with the Declaration of Helsinki and International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use Guideline for Good Clinical Practice guidelines. The protocol has been approved by the institutional review board of the lead institution and by ethics committees at all participating sites. Written informed consent will be obtained from all participants before any study-specific procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed small bowel adenocarcinoma (duodenum excluding the ampulla of Vater, jejunum, or ileum). If pathology was performed at another institution, slides/blocks must be reviewed by a pathologist at the study site before enrollment.
2. One of the following:

   1. unresectable locally advanced small bowel adenocarcinoma in which R0 resection would require combined resection of invaded organs and is judged infeasible
   2. UICC-TNM stage IV small bowel adenocarcinoma with distant metastasis
   3. postoperative recurrence of small bowel adenocarcinoma.
3. No symptomatic brain metastases, carcinomatous meningitis, or spinal metastases requiring radiation or surgical intervention.
4. No clinically significant pericardial effusion, pleural effusion, or ascites requiring treatment.
5. Age ≥18 years at registration.
6. Eastern Cooperative Oncology Group performance status (ECOG PS) 0-1.
7. ≥1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1, on contrast-enhanced CT (slice thickness ≤5 mm) obtained within 14 days before registration.
8. Prior platinum-based chemotherapy for unresectable locally advanced or metastatic small bowel adenocarcinoma (FOLFOX or CapeOX) with documented progression, recurrence or treatment discontinuation due to toxicity.
9. If prior testing (e.g., microsatellite instability, mismatch repair, or comprehensive genomic profiling) has identified alterations that qualify for tumor-agnostic approved therapies, the patient must be refractory, intolerant, or ineligible to such therapies. These tests are not mandatory; lack of testing does not preclude enrollment.
10. Archival tumor tissue is available; if unavailable, the patient agrees to a pre-treatment biopsy to obtain tumor tissue.
11. No anticancer chemotherapy or radiotherapy within 14 days before registration.
12. No surgery under general anesthesia within 28 days before registration.
13. Screening laboratory tests within 14 days before registration meet all of the following conditions:

    1. absolute neutrophil count ≥1,500/mm³
    2. platelet count≥100,000/mm³
    3. hemoglobin ≥8.5 g/dL
    4. AST ≤100 U/L (≤200 U/L with liver metastases)
    5. ALT ≤100 U/L (≤200 U/L with liver metastases)
    6. total bilirubin ≤1.5 mg/dL
    7. serum creatinine ≤1.5 mg/dL
14. Contraception: Women of childbearing potential agree to use effective contraception and to refrain from oocyte donation from consent through ≥2 months after last dose; breastfeeding patients agree to withhold breastfeeding for ≥3 weeks after last dose; men agree to use effective contraception and to refrain from sperm donation from consent until ≥1 month after last dose.
15. Written informed consent obtained from the patient.

Exclusion Criteria:

1. Active second primary malignancy.
2. Active infection requiring systemic therapy.
3. Interstitial lung disease/pneumonitis, diagnosed by imaging or clinical findings, current or prior, irrespective of steroid use.
4. Poorly controlled diabetes mellitus: HbA1c ≥8%, or HbA1c 7.0-<8.0% with otherwise unexplained hyperglycemic symptoms (polyuria and/or polydipsia).
5. Known hypersensitivity to enfortumab vedotin, its excipients (e.g., histidine, trehalose dihydrate, polysorbate 20).
6. Ongoing grade ≥2 sensory or motor peripheral neuropathy.
7. Cerebrovascular event, unstable angina, myocardial infarction, or severe heart failure within 6 months before registration.
8. Ongoing grade ≥2 unresolved clinically significant toxicities from prior therapy, excluding alopecia.
9. Ongoing grade ≥2 dermatologic disorders regardless of prior-treatment causality.
10. Ongoing use of chronic systemic corticosteroids or other immunosuppressants.
11. Active keratitis or corneal ulcer.
12. Positive for HIV antibodies, HBs antigen, or HCV RNA
13. Negative for HBs antigen, positive for HBs or HBc antibodies, and positive HBV DNA quantification (patients are not excluded if HBV DNA is detected but below the limit of quantification).
14. Pregnant or possibly pregnant women.
15. Psychiatric illness or psychiatric symptoms that interfere with activities of daily living and, in the investigator's judgment, preclude study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate by central review | Overall response will be assessed every 8 weeks through 24 weeks, then every 12 weeks thereafter, from baseline up to 3 years or until disease progression or post-study treatment, whichever occurs first.
  The objective response rate is defined as the proportion of patients in the full analysis set whose best overall response is a complete response (CR) or partial response (PR). Best overall response is defined as the best response recorded among CR, PR, stable disease (SD), progressive disease (PD), and not evaluable (NE) using RECIST version 1.1.

SECONDARY OUTCOMES:
Objective response rate by institutional review | Overall response will be assessed every 8 weeks through 24 weeks, then every 12 weeks thereafter, from baseline up to 3 years or until disease progression or post-study treatment, whichever occurs first.
  Objective response rate is defined as the proportion of patients in the full analysis set whose best overall response is a complete response (CR) or partial response (PR). Best overall response is defined as the best response recorded among CR, PR, stable disease (SD), progressive disease (PD), and not evaluable (NE) using RECIST version 1.1.
Progression-free survival | From baseline up to 3 years
  Progression-free survival for each participant in the full analysis set is defined as the period from the date of enrollment to the date on which PD is confirmed by institutional review or the date of death from any cause, whichever comes first.
Overall survival | From baseline up to 3 years
  Overall survival for each participant in the full analysis set is defined as the period from the date of enrollment to the date of death from any cause.
Disease control rate | From baseline up to 3 years
  Disease control rate is defined as the percentage of participants in the full analysis set with the best overall response of CR, PR, and SD. The disease control rate is calculated based on both institutional review and central review.
Incidence of adverse events | From baseline up to 3 years
  Incidence of adverse events is defined as the percentage of participants in the safety analysis set who experienced each adverse event. In addition, the frequency of the worst grade by CTCAE v5.0-JCOG will be calculated for each adverse event.
Dose Intensity | From baseline up to 3 years
  Dose Intensity is calculated for each participant as the actual total dose of the study drug administered from the start of treatment to the last dose, normalized by the participant's body weight at enrollment, divided by the treatment duration in weeks.
Relative dose intensity | From baseline up to 3 years
  Dose Intensity is calculated for each participant as the actual total dose of the study drug administered from the start of treatment to the last dose, normalized by the participant's body weight at enrollment, divided by the treatment duration in weeks.
Duration of response | From baseline up to 3 years
  Duration of response for each participant in the full analysis set is defined as the period from the date on which CR or PR is first confirmed to the date on which PD is confirmed by institutional review or the date of death from any cause, whichever comes first.
Time to response | From baseline up to 3 years
  Time to response for each participant in the full analysis set is defined as the period from the date of enrollment to the date on which CR or PR is first confirmed based on both institutional review and central review.

OTHER OUTCOMES:
Objective response rate according to Nectin-4 expression status | Overall response will be assessed every 8 weeks through 24 weeks, then every 12 weeks thereafter, from baseline up to 3 years or until disease progression or post-study treatment, whichever occurs first.
  A subgroup analysis of the objective response rate is conducted according to Nectin-4 expression status at baseline.Nectin-4 expression is assessed on a scale of 0 to 3.

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Kyushu University Hospital, Fukuoka
  - Osaka International Cancer Institute, Osaka
  - National Cancer Center Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fujii H, Shoji H, Hirano H, Hirose T, Okita N, Takashima A, Kato K. Exploring novel therapeutic targets in small bowel adenocarcinoma: insights from claudin 18.2, nectin-4, and HER3 expression analysis. ESMO Open. 2025 Jan;10(1):104098. doi: 10.1016/j.esmoop.2024.104098. Epub 2025 Jan 3. PMID 39754977